CLINICAL TRIAL: NCT02071823
Title: Single Dose Crossover Comparative Bioavailability Study of BIA 9-1067 25 mg Capsules in Healthy Male Volunteers Following Administration of a 50 mg Dose / Fasted and Fed States
Brief Title: Comparative Bioavailability Study of BIA 9-1067 25 mg Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-104
Record Dates: First submitted 2012-01-19; First posted 2014-02-26 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2014-12

CONDITIONS: Parkinson
Keywords: Opicapone,; Parkinson,; Bial,; BIA 9-1067
MeSH Terms: interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A Fed/Fasted (Experimental): A single 50 mg dose of BIA 9-1067 (2 x 25 mg capsules) was to be administered on:
  Period 1: Fed Washout Period (7days) Period 2: Fasted
  Interventions: Drug: BIA 9-1067
- Group B Fasted/Fed (Experimental): A single 50 mg dose of BIA 9-1067 (2 x 25 mg capsules) was to be administered on:
  Period 1: Fasted Washout Period (7days) Period 2: Fed
  Interventions: Drug: BIA 9-1067

INTERVENTIONS:
Drug: BIA 9-1067 — A single oral dose of 50 mg (2 x 25 mg capsules) was administered in the morning of each study period under fasting or fed conditions. The two single dose administrations were separated by a wash-out of 7 days.
  Other Names: Opicapone, OPC

SUMMARY:
The objectives of this study were to characterize the effects of food on the pharmacokinetics (PK) and tolerability of BIA 9-1067 in healthy male subjects.

DETAILED DESCRIPTION:
Methodology: Single center, randomized, single dose, open-label, 2-period, 2-sequence, crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Availability for the entire study period and willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read, signed and dated by the volunteer
* Male volunteer
* Volunteer aged of at least 18 years but not older than 45 years
* Volunteer with a body mass index (BMI) greater than or equal to 18.5 and below 30 kg/m2
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance
* Healthy according to the medical history, laboratory results and physical examination
* Light-, non- or ex-smokers. A light smoker is defined as someone smoking 10 cigarettes or less per day for at least 3 months before day 1 of this study. An ex-smoker is defined as someone who completely stopped smoking for at least 12 months before day 1 of this study
* The informed consent form must be signed by all volunteers, prior to their participation in the study.

Exclusion Criteria:

* Volunteers presenting any of the following will not be included in the study:Significant history of hypersensitivity to any catechol-structured drugs (e.g. rimiterole, isoprenaline, adrenaline, noradrenaline, dopamine, dopexamine or dobutamide) or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
* Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic, dermatologic or connective tissue disease
* Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
* Presence of significant heart disease or disorder according to ECG
* Previous history of Neuroleptic Malignant Syndrome (NMS) and/or nontraumatic rhabdomyolysis
* Pheochromocytoma due to the increased risk of hypertensive crisis
* Use of MAO inhibitors within 14 days of day 1 of the study
* Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin and rifampin), in the previous 28 days before day 1 of this study
* Volunteers who took an Investigational Product (in another clinical trial) or donated 50 mL or more of blood in the previous 28 days before day 1 of this study
* Poor motivation, intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with the protocol requirements or inability to cooperate adequately, inability to understand and to observe the instructions of the physician
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study
* Positive urine screening of drugs of abuse
* Any history of tuberculosis and/or prophylaxis for tuberculosis
* Positive results to HIV, HBsAg or anti-HCV tests

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A Fed/Fasted: A single 50 mg dose of BIA 9-1067 (2 x 25 mg capsules) was to be administered on:
  Period 1: Fed Washout Period (7days) Period 2: Fasted
  BIA 9-1067: A single oral dose of 50 mg (2 x 25 mg capsules) was administered in the morning of each study period under fasting or fed conditions. The two single dose administrations were separated by a wash-out of 7 days.
- Group B Fasted/Fed: A single 50 mg dose of BIA 9-1067 (2 x 25 mg capsules) was to be administered on:
  Period 1: Fasted Washout Period (7days) Period 2: Fed
  BIA 9-1067: A single oral dose of 50 mg (2 x 25 mg capsules) was administered in the morning of each study period under fasting or fed conditions. The two single dose administrations were separated by a wash-out of 7 days.
Period: Overall Study
Arm/Group | Group A Fed/Fasted | Group B Fasted/Fed
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A Fed/Fasted | Group B Fasted/Fed | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Description: Cmax - Maximum observed plasma concentration of BIA 9-1067
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fasted Conditions: Fasted conditions period
- Fed Condition: Fed condition period
Arm/Group | Fasted Conditions | Fed Condition
Number analyzed (Participants) | 11 | 11
ng/mL | 635.0 (250.8) | 238.2 (168.4)

2. Primary Outcome: AUCt - Cumulative Area Under the Plasma Concentration Time Curve
Description: AUCt - Cumulative Area Under the plasma concentration time Curve for BIA 9-1067
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng·h/mL
Groups:
- Fed Conditions: Fed conditions period
- Fasted Condition: Fasted condition period
Arm/Group | Fed Conditions | Fasted Condition
Number analyzed (Participants) | 11 | 11
ng·h/mL | 879.2 (286.6) | 1989.5 (984.8)

3. Primary Outcome: Area Under the Concentration-time Curve Extrapolated to Infinity (AUC∞)
Description: Area Under the Concentration-time Curve Extrapolated to Infinity (AUC∞) for BIA 9-1067
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Fasted Conditions | Fed Condition
Number analyzed (Participants) | 11 | 11
ng·h/mL | 2113.6 (915.2) | 1027.2 (545.4)

ADVERSE EVENTS:
Arm/Group | Fasted Conditions | Fed Condition
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 3/11 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fasted Conditions (N=11) | Fed Condition (N=12)
Somnolence (Nervous system disorders) | 2 | 4
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other